CLINICAL TRIAL: NCT00080496
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Comparative Study Of The Efficacy And Safety Of Tigecycline Vs Imipenem/Cilastatin For The Treatment Of Subjects With Nosocomial Pneumonia
Brief Title: Study Evaluating Tigecycline Versus Imipenem/Cilastatin in Hospital-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3074A1-311
Record Dates: First submitted 2004-04-05; First posted 2004-04-07 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-07

CONDITIONS: Bacterial Pneumonia
Keywords: Pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia | interventions — Tigecycline; Imipenem; Cilastatin

INTERVENTIONS:
Drug: Tigecycline
Drug: Imipenem
Drug: Cilastatin

SUMMARY:
To compare the efficacy and safety of the tigecycline regimen with that of the imipenem/cilastatin regimen in subjects with nosocomial pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over 18 years of age. Bulgaria Only: Male or female subjects over 18 years of age and under 70 years of age.
* Subjects known or suspected to have acute hospital-acquired pneumonia.

Exclusion Criteria:

* Presence of any of the following pulmonary conditions: cystic fibrosis; pulmonary malignancy (either primary or metastatic); known bronchial-obstructive or post obstructive pneumonia; pulmonary abscess; empyema; known or suspected active tuberculosis; bronchiectasis; sarcoidosis; known or suspected pulmonary infection caused by Pneumocystis carinii, mycobacteria, fungi, parasites, or viruses (Subjects with COPD are not excluded)
* Suspected or known Legionella infection
* Concurrent hemodialysis, hemofiltration, peritoneal dialysis, or plasmapheresis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430
Dates: Start 2003-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The co-primary efficacy endpoints are clinical response at the TOC assessment for the clinically evaluable population and the clinical modified intent-to-treat population.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (24):
- United States (24):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Martinez, California
  - Modesto, California
  - National City, California
  - Bay Pines, Florida
  - Crystal River, Florida
  - Gainesville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Roswell, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Columbia, Missouri
  - Omaha, Nebraska
  - Henderson, North Carolina
  - Cincinnati, Ohio
  - Zanesville, Ohio
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina

REFERENCES:
- [Derived] Karageorgopoulos DE, Kelesidis T, Kelesidis I, Falagas ME. Tigecycline for the treatment of multidrug-resistant (including carbapenem-resistant) Acinetobacter infections: a review of the scientific evidence. J Antimicrob Chemother. 2008 Jul;62(1):45-55. doi: 10.1093/jac/dkn165. Epub 2008 Apr 24. PMID 18436554